CLINICAL TRIAL: NCT05589376
Title: You and Me Healthy Registry Study
Brief Title: You and Me Healthy
Acronym: YMH
Status: Enrolling by invitation | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00110716
Record Dates: First submitted 2022-09-28; First posted 2022-10-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The You and Me Healthy Registry provides a resource for collecting information on people currently living in the United States. The overall goal of the Registry is to create and engage a community of people who may be eligible for participation in future research studies aiming to answer research questions about COVID-19 and other conditions.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a novel betacoronavirus responsible for the COVID-19 pandemic. In the United States (US) up until January 2022, > 60 million people have been infected with the SARS-CoV-2 virus and >800,000 died, with infections and deaths disproportionally affecting populations that have been historically marginalized1. Wide disparities also persist by race/ethnicity and age with COVID-19 testing and vaccine uptake related to social and structural factors, resulting in adverse health consequences.

As public health measures have scaled up, mitigation strategies are increasingly being considered to reduce community spread of infection. These measures include rapid-result at-home tests, protective measures (masking, social distancing, increased hygiene), treatments, and contact-tracing and isolation. As the pandemic evolves, new discoveries, technologies, and strategies to combat COVID-19 are being implemented with limited backing of research data. To address this continued unmet public health need, the You and Me Healthy registry is being created to engage community members and serve as a way to provide and collect information from all people who are interested in engaging in upcoming research studies, including those related to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Currently residing in the United States
* Age ≥ 2 (for minors, parents/legal guardian will be the primary point of contact)
* Able to speak and read in the language used in the surveys/assessments available

Exclusion Criteria:

There are no specific exclusion criteria for this registry

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The You and Me Healthy Registry will include children and adults currently living across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants enrolled in the Virtual Community | Through study completion; 5 years
  Create a virtual community of people in the United States interested in engaging in upcoming research studies, including those related to COVID-19; By asking them to sign -up and join the registry- they provide their email address and through that they will receive information on upcoming research and information on health issues occurring in their community.
Number of participants included in the Dataset | Through study completion; 5 years
  Create a dataset of health-related measurements, risk factors, and outcomes for future; analysis and in support of upcoming research studies; through collecting survey responses via questioners.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hornik, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Merced County, Merced, California
  - Greenville Pitt County, Greenville, North Carolina
  - Hamilton County, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Agostino EM, Granados I, Abbott-Grimes P, Brown-Lowery C, Damman A, Fadika T, Ward M, Cooper M, Sato J, Kasper J, Vizcaino T, Gray W, Swart A, Sparling A, Corchado CG, Hornik CP. Community partnership lessons learned from the You & Me: Test and Treat study. BMC Public Health. 2025 Jun 6;25(1):2115. doi: 10.1186/s12889-025-23216-y. PMID 40481451